CLINICAL TRIAL: NCT01210651
Title: Treating Major Depression With Yoga: A Prospective, Randomized Controlled Pilot Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Mental Insight Foundation (Unknown); Pritzker Family Foundation (Other); Mount Zion Health Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H49362-35940-01
Record Dates: First submitted 2010-09-21; First posted 2010-09-28 (Estimated); Results first posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Depression, Unipolar
Keywords: Yoga; Major Depression; Self-Efficacy; Self-Esteem; Hatha yoga; mind-body therapies; depression
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hatha Yoga Practice Group (Experimental): Participants in this group practiced 90-minute sessions of hatha yoga exercises twice weekly for a total of 8 weeks.
  Interventions: Behavioral: Hatha Yoga Practice Group
- Attention Control Education Group (Active Comparator): Participants in this group attended 90-minute educational seminars on yoga history twice weekly for a total of 8 weeks.
  Interventions: Behavioral: Attention Control Education Group

INTERVENTIONS:
Behavioral: Hatha Yoga Practice Group — The hatha yoga intervention was a sequence of classical yoga practices, comprised of breathing techniques, mindful body postures, and a final deep relaxation pose. The same sequence was used in all sessions. Yoga practices were broken down into component elements and taught progressively to each student in accordance with his or her ability. Participants were encouraged to remain within their range of motion or comfort. Accommodations were made for those with limitations in tolerance or flexibility for any exercise. Blocks, bolsters and other props were used to support participants in learning and holding yoga poses safely, particularly during back-bends or inverted poses. The intervention was delivered by a licensed, registered nurse, who was also a registered yoga teacher.
  Other Names: Yoga Practice Group, Hatha Yoga Group, Yoga Exercise Group
  Arms: Hatha Yoga Practice Group
Behavioral: Attention Control Education Group — The educational seminars taught to participants covered the history and philosophy of the main branches of yoga. Documentary films were used during the seminars to enhance lectures, and interactive dialogue was encouraged between instructor and participants. Seminars were designed to control for non-specific mood benefits of study participation, such as attention from instructors, peer interaction, time spent away from routine activities, and anticipation/interest related to mastering novel yoga-related information. Since participants would join the attention control group on a rolling basis, seminars were designed to function as stand-alone educational modules, rather than requiring presentation in a specific sequence. The instructor for the seminars was a registered yoga teacher.
  Other Names: Attention Control Group, Education Group, Yoga History Group
  Arms: Attention Control Education Group

SUMMARY:
This was a randomized controlled pilot trial to evaluate clinical efficacy and feasibility of hatha yoga as a mono-therapy for major depression. Investigators recruited 38 adults in San Francisco meeting criteria for major depression of mild-to-moderate severity, per structured psychiatric interview and scores of 14-28 on Beck Depression Inventory-II (BDI). At screening, individuals engaged in psychotherapy, antidepressant pharmacotherapy, herbal/nutraceutical mood therapies, or mind-body practices were excluded. Twenty participants were randomized to 90-minute hatha yoga practice groups twice weekly for 8 weeks. Eighteen participants were randomized to 90-minute attention control education groups twice weekly for 8 weeks. Certified yoga instructors delivered both interventions at a university clinic. Primary outcome was depression severity, measured by BDI scores every 2 weeks from intervention start at 0 weeks until finish at 8 weeks. Secondary outcomes were self-efficacy and self-esteem, measured by scores on the General Self-Efficacy Scale (GSES) and Rosenberg Self-Esteem Scale (RSES) at 0 weeks and 8 weeks. Blinded assessors analyzed whether change in outcome measures would be statistically comparable between the two intervention groups.

DETAILED DESCRIPTION:
This was a prospective, single-center, single-blind, randomized, controlled, parallel group, pilot trial of an 8-week hatha yoga program as mono-therapy in major depression. Recruitment occurred from May to October 2010, and the trial was concluded in January 2011.

We recruited 38 adults from the San Francisco community who met criteria for major depression of mild-to-moderate severity, as per screening diagnostic evaluation with the Mini International Neuropsychiatric Interview (MINI) and scores of 14 through 28 on the Beck Depression Inventory-II (BDI). At screening, individuals engaged in psychotherapy, antidepressant pharmacotherapy, herbal/nutraceutical mood remedies, or any mind-body practices were excluded.

Eligible participants were randomized in a 1:1 ratio to one of two instructor-led intervention groups: a hatha yoga practice group assigned to 90-minute hatha yoga practice sessions twice weekly for 8 weeks, versus an attention control education group assigned to 90-minute yoga history seminars twice weekly for 8 weeks. Participants in the hatha yoga group learned and practiced a specific sequence of classical yoga breathing techniques, mindful body postures, and a final deep relaxation pose. The attention control education group explored the history and philosophy of the main branches of yoga through seminars featuring lectures, documentary films, and interactive dialogue between instructor and participants; the seminars were designed to control for non-specific mood benefits of the hatha yoga intervention, such as attention from study personnel, peer interaction, time spent away from routine activities, and anticipation/interest related to mastering novel yoga-related information.

Stratified block randomization was undertaken to ensure that each intervention group had equal numbers of participants with mild depression (per screening BDI scores of 14 to 19) versus moderate depression (per screening BDI scores of 20 to 28).

Participants were informed at screening that anyone randomized to the education group would be offered 16 free hatha yoga classes, upon completion of the study, to learn and practice the same exercises taught to the hatha yoga practice group.

The primary outcome was depression severity, measured by BDI scores at 2-week intervals from intervention start at 0 weeks until intervention end at 8 weeks. Secondary outcomes were self-efficacy and self-esteem, measured respectively by scores on the General Self-Efficacy Scale (GSES) and the Rosenberg Self-Esteem Scale (RSES) at 0 weeks and at 8 weeks. Blinded assessors analyzed outcome data from both intervention groups, testing whether change in outcome measures would be statistically comparable between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 14 years of age and older
* English proficiency sufficient for study participation
* Diagnosis of Axis I unipolar major depression, per screening Mini International Neuro-Psychiatric Interview (MINI)
* Depressive symptoms of mild to moderate intensity, per score of 14-28 on screening Beck Depression Inventory-II (BDI)
* Able to attend all required study sessions

Exclusion Criteria:

* Cognitive Impairment, as per Folstein Mini-mental Status Exam Score < 24
* Use of any antidepressant medication or herbal/nutraceutical mood therapy within the 2 months prior to screening, or during study period
* Use of psychotherapy during study period
* Use of any yoga or other mind-body practices during study period, other than study intervention
* Per screening MINI, diagnosis of any Axis I disorder other than unipolar major depression, such as bipolar disorder, dysthymia or anxiety disorders
* Per screening MINI, diagnosis of substance use disorders within prior 3 months
* Per screening MINI, current suicidal ideation or past suicide attempts
* Severe depressive symptoms, as per screening BDI score > 28

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudha Prathikanti, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data from this clinical trial have been de-identified of any protected health information, and made available for sharing with other researchers. The dataset includes demographic/clinical variables obtained from all randomized participants at screening, as well as primary and secondary outcome measures obtained from participants in both intervention groups over the course of the 8-week intervention period. The dataset is accessible as an Excel file via the following web link: http://prathikanti.com/studydata/

REFERENCES:
- [Derived] Prathikanti S, Rivera R, Cochran A, Tungol JG, Fayazmanesh N, Weinmann E. Treating major depression with yoga: A prospective, randomized, controlled pilot trial. PLoS One. 2017 Mar 16;12(3):e0173869. doi: 10.1371/journal.pone.0173869. eCollection 2017. PMID 28301561

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via consecutive sampling of eligible individuals responding to ads approved by the Institutional Review Board of the University of California, San Francisco. Ads were posted in San Francisco libraries, shopping areas, community centers, outpatient clinics, local newspapers, online classifieds & clinical trials websites.
Groups:
- Hatha Yoga Practice Group: Participants in this group met for 90-minute yoga practice sessions twice a weekly for a total of 8 weeks.
- Attention Control Education Group: Participants in this group met for 90-minute educational seminars on yoga history twice weekly for a total of 8 weeks.
Period: Overall Study
Arm/Group | Hatha Yoga Practice Group | Attention Control Education Group
Started | 20 (Number randomized to intervention, but not number who started intervention by attending 1st session.) | 18 (Number randomized to intervention, but not number who started intervention by attending 1st session.)
Number Attending 1st Assigned Session | 18 | 12
Completed | 15 | 10
Not Completed | 5 | 8
Not completed — Lost to Follow-up | 1 | 1
Not completed — schedule conflicts | 1 | 5
Not completed — Withdrawn by PI for disruptive behavior | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Injury outside study | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population comprised of all participants randomized to the 2 intervention groups, regardless of whether participants subsequently began intervention by attending the first assigned session at 0 weeks.
Groups:
- Hatha Yoga Practice Group: Participants in this group met for 90-minute sessions of hatha yoga practice twice a week for a total of 8 weeks.
- Attention Control Education Group: Participants in this group met for 90-minute education seminars on yoga history twice a week for a total of 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Hatha Yoga Practice Group | Attention Control Education Group | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] — Participant provided birthdate at the time of the office screening visit, and age was calculated as of the screening date.
  years | 43.1 (15.2) | 43.8 (14.7) | 43.4 (14.8)
Age, Customized [Number; unit: years] — Age range of participants, with ages calculated as of the screening visit date.
  years
    Lowest age among participants | 22 | 23 | 22
    Highest age among participants | 64 | 72 | 72
Gender [Count of Participants; unit: Participants]
  Female | 15 | 11 | 26
  Male | 5 | 7 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participant provided self-described ethnic identity at the time of the office screening visit.
  Participants
    European descent | 13 | 9 | 22
    Asian descent | 2 | 4 | 6
    Latino descent | 2 | 2 | 4
    African descent | 1 | 2 | 3
    Multi-ethnic descent | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 20 | 18 | 38
Married [Count of Participants; unit: Participants] — Participant provided information on marital status at the time of the office screening visit.
  Participants | 1 | 3 | 4
Highest Education [Count of Participants; unit: Participants] — Participant provided information on highest level of education attained at the time of the office screening visit.
  Participants
    High school diploma | 0 | 2 | 2
    Two years of college | 5 | 7 | 12
    Four-year college degree or higher | 15 | 9 | 24
Employment [Count of Participants; unit: Participants]
  Employed | 8 | 12 | 20
  Student | 2 | 2 | 4
  Retired | 3 | 2 | 5
  Unemployed | 7 | 2 | 9
Prior Yoga Exposure [Count of Participants; unit: Participants] — Prior yoga exposure was defined as the report during screening of any past participation in any individual or group yoga classes/exercises.
  Participants | 10 | 14 | 24
Participants with Prior Depressive Episodes [Count of Participants; unit: Participants] — During the Mini International Neuro-Psychiatric Interview conducted at screening, participant was asked questions to ascertain the number of any prior discrete mood episodes meeting criteria for unipolar major depression.
  Participants
    Participants with 0 prior episodes | 3 | 1 | 4
    Participants with 1 prior episode | 12 | 10 | 22
    Participants with 2 prior episodes | 4 | 5 | 9
    Participants with 3 prior episodes | 1 | 2 | 3
Participants with Prior Antidepressant Trials [Count of Participants; unit: Participants] — During the Mini International Neuro-Psychiatric Interview conducted at screening, participant reported on the total number of anti-depressant medication trials, if any, received as treatment during any prior depressive episodes.
  Participants
    Participants with 0 prior trials | 10 | 3 | 13
    Participants with 1 prior trial | 5 | 10 | 15
    Participants with 2 prior trials | 2 | 3 | 5
    Participants with 3 prior trials | 3 | 1 | 4
    Participants with 4+ prior trials | 0 | 1 | 1
Screening Score on Beck Depression Inventory-II [Mean (Standard Deviation); unit: points on a scale] — The Beck Depression Inventory-II (BDI) is a 21-item validated instrument for the self-report of depressive symptoms, with individual item scores summed to yield a total possible BDI score that ranges from 0-63. BDI scores from 0-13 suggest absent to minimal depressive symptoms, from 14-19 mild symptoms, from 20-28 moderate symptoms, and from 29-63 severe symptoms.
  points on a scale | 22.8 (4.4) | 22.4 (4.6) | 22.4 (4.5)
Screening Score on Folstein Mini Mental Status Exam [Mean (Standard Deviation); unit: points on a scale] — The Folstein Mini Mental Status Exam (MMSE) is a validated, clinician-administered instrument for assessing cognition via tests of orientation, attention, calculation, memory, and both written and spoken language. Scores from each cognitive test are summed to derive a total score ranging from 0 (worst score) to 30 (best score). Cognitive performance as measured by the MMSE varies within the population by age and educational level, but scores below 24 may suggest cognitive impairment.
  points on a scale | 27.7 (1.8) | 28.4 (1.2) | 28.0 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Intent-to-Treat Analysis of Adjusted Mean Beck Depression Inventory-II Scores Over Intervention Period
Description: The Beck Depression Inventory-II (BDI) is a 21-item validated instrument for the self-report of depressive symptoms, with individual item scores summed to yield a total possible BDI score that ranges from 0-63. BDI scores from 0-13 suggest absent to minimal depressive symptoms, from 14-19 mild symptoms, from 20-28 moderate symptoms, and from 29-63 severe symptoms. Regression analysis software examined the BDI scores measured in study participants every 2 wks from intervention start at 0 wks until intervention end at 8 wks, using maximum likelihood estimations to derive an adjusted mean BDI score for each intervention group at each measurement point.
Time Frame: 0 wks, 2 wks, 4 wks, 6 wks, 8 wks
Population: Intent-to-Treat population was comprised of all randomized participants in both intervention groups, regardless of adherence to protocol or premature dropout. BDI scores of any participants missing at 0 wks were imputed by carrying forward their BDI scores from screening.
Measure: Least Squares Mean (95% Confidence Interval); unit: points on a scale
Arm/Group | Hatha Yoga Practice Group | Attention Control Education Group
Number analyzed (Participants) | 20 | 18
points on a scale
  Adjusted Mean BDI Score at 0 wks | 20.98 [18.45 to 23.51] | 19.92 [17.26 to 22.58]
  Adjusted Mean BDI Score at 2 wks | 15.15 [12.17 to 18.12] | 13.06 [8.91 to 17.20]
  Adjusted Mean BDI Score at 4 wks | 14.35 [11.28 to 17.41] | 14.66 [10.76 to 18.56]
  Adjusted Mean BDI Score at 6 wks | 13.04 [9.46 to 16.62] | 12.72 [7.82 to 17.62]
  Adjusted Mean BDI Score at 8 wks | 11.51 [8.69 to 14.33] | 16.93 [13.56 to 20.30]
Statistical Analysis 1: Comparison: Hatha Yoga Practice Group vs Attention Control Education Group; A random-effects, generalized least squares (GLS) regression model for depression severity was used to analyze participant BDI scores measured just before 1st assigned session at 0 wks, and just after assigned sessions at 2 wks, 4 wks, 6 wks and 8 wks. BDI Scores were modeled as correlated within participants but independent between participants. The GLS regression model tested the null hypothesis that no significant effects on BDI scores would be found by intervention and intervention-by-time; Test type: Superiority or Other; p = 0.034, Regression, Generalized Least Squares — Analysis performed via Stata v14.1. Alpha was 2-tailed. P-value was calculated, with p-value < 0.05 required a priori to reject the null hypothesis

2. Primary Outcome: Total Change Scores on Beck Depression Inventory-II Among Study Completers
Description: The Beck Depression Inventory-II (BDI) is a 21-item validated instrument for the self-report of depressive symptoms, with individual item scores summed to yield a total possible BDI score that ranges from 0-63. BDI scores from 0-13 suggest absent to minimal depressive symptoms, from 14-19 mild symptoms, from 20-28 moderate symptoms, and from 29-63 severe symptoms. BDI scores of study completers were examined, and the total change score on BDI was calculated for each intervention group as the mean BDI score at 0 wks subtracted from the mean BDI score at 8 wks.
Time Frame: 0 wks and 8 wks
Population: Population of study completers was comprised of participants in both intervention groups who provided study measures at intervention start at 0 wks and at intervention end at 8 wks.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Hatha Yoga Practice Group | Attention Control Education Group
Number analyzed (Participants) | 15 | 10
points on a scale
  Mean BDI Score at 0 wks | 20.47 (6.00) | 18.00 (6.43)
  Mean BDI Score at 8 wks | 11.00 (10.01) | 16.30 (7.63)
  Total Change Score on BDI | -9.47 (8.85) | -1.70 (6.67)
Statistical Analysis 1: Comparison: Hatha Yoga Practice Group vs Attention Control Education Group; Statistical analysis examined Total Change Scores on BDI, using two sample t-test to evaluate the null hypothesis that the Total Change Score on BDI for each intervention group would be statistically comparable; Test type: Superiority or Other; p = 0.02, t-test, 2 sided — Analysis performed via Stata v14.1, with P-value calculated using a t-distribution and assuming unequal variances in the two samples. Alpha was two-tailed. P-value < 0.05 was required a priori to reject the null hypothesis

3. Primary Outcome: Number of Study Completers With Remitted Depression, Per Completers Analysis of BDI Scores at 8 Weeks
Description: The Beck Depression Inventory-II (BDI) is a 21-item validated instrument for the self-report of depressive symptoms, with individual item scores summed to yield a total possible BDI score that ranges from 0-63. BDI scores from 0-13 suggest absent to minimal depressive symptoms, from 14-19 mild symptoms, from 20-28 moderate symptoms, and from 29-63 severe symptoms. Analysis examined BDI scores of study completers and identified in each intervention group the number of participants with an 8-wk BDI score ≤ 9, defined as remitted depression.
Time Frame: 8 Weeks
Population: Population of study completers with remitted depression was comprised of participants in both intervention groups who provided study measures at 0 wks and 8 wks, and achieved an 8-wk BDI score ≤ 9.
Measure: Number; unit: participants
Groups:
- Attention Control Education Group: Participants in this group met for 90-minute educational seminars on yoga history twice a week for a total of 8 weeks.
Arm/Group | Hatha Yoga Practice Group | Attention Control Education Group
Number analyzed (Participants) | 15 | 10
participants
  Number of Study Completers with 8-wk BDI score ≤ 9 | 9 | 1
  Number of Study Completers with 8-wk BDI score > 9 | 6 | 9
Statistical Analysis 1: Comparison: Hatha Yoga Practice Group vs Attention Control Education Group; Fisher's Exact test evaluated null hypothesis that the proportion of study completers with remitted depression would be statistically comparable in the 2 intervention groups; Test type: Superiority or Other; p = 0.018, Fisher Exact — Analysis performed via Stata v14.1. Alpha was 2-tailed. P-value was calculated, with a p-value < 0.05 required a priori to reject the null hypothesis

4. Secondary Outcome: Total Change Scores on General Self-Efficacy Scale (GSES) Among Study Completers
Description: The General Self-Efficacy Scale (GSES) is a 10-item, self-administered, validated psychometric instrument to measure self-efficacy, defined as the belief that one's actions are responsible for successful outcomes in coping with difficult life demands. Each item is scored from 1 to 4, with a total GSES score derived by summing the individual item scores. Possible GSES scores range from 10 (no belief in one's self-efficacy) to 40 (strongest belief in one's self-efficacy). GSES scores of study completers were examined, and the total change score on GSES was calculated for each intervention group as the mean GSES score at 0 wks subtracted from the mean GSES score at 8 wks.
Time Frame: 0 wks, 8 wks
Population: Population of study completers was comprised of participants in both intervention groups who provided study measures at intervention start at 0 wks and at intervention finish at 8 wks.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Hatha Yoga Practice Group | Attention Control Education Group
Number analyzed (Participants) | 15 | 10
points on a scale
  Mean GSES Score at 0 wks | 26.87 (3.09) | 28.50 (4.33)
  Mean GSES Score at 8 wks | 29.00 (3.89) | 30.00 (2.67)
  Total Change Score on GSES | 2.13 (2.07) | 1.50 (2.37)
Statistical Analysis 1: Comparison: Hatha Yoga Practice Group vs Attention Control Education Group; Statistical analysis examined Total Change Scores on GSES, using an independent samples t-test to evaluate null hypothesis that Total Change Score on GSES for each intervention group would be statistically comparable; Test type: Superiority or Other; p = 0.50, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]

5. Secondary Outcome: Total Change Scores on Rosenberg Self-Esteem Scale (RSES) Among Study Completers
Description: The Rosenberg Self-Esteem Scale (RSES) is a 10-item, self-administered, validated psychometric instrument to measure self-esteem, defined as having an overall feeling of self-worth and self-acceptance. Each item is scored from 0 to 3, and individual item scores are summed to yield a total possible RSES ranging from 0-30. RSES scores from 0-14 suggest low self-esteem, from 15-25 normal self-esteem, and from 26-30 high self-esteem. RSES scores of study completers were examined, and the total change score on RSES was calculated for each intervention group as the mean RSES score at 0 wks subtracted from the mean RSES score at 8 wks.
Time Frame: 0 wks, 8 wks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: points on a scale
Groups:
- Yoga Practice Group: Participants in this group met for 90-minute sessions of hatha yoga practice twice a week for a total of 8 weeks.
- Attention Control Group: Participants in this group met for 90-minute educational seminars on yoga history twice a week for a total of 8 weeks.
Arm/Group | Yoga Practice Group | Attention Control Group
Number analyzed (Participants) | 15 | 10
points on a scale
  Mean RSES Score at 0 wks | 14.6 (3.48) | 16.0 (3.77)
  Mean RSES Score at 8 wks | 17.47 (3.87) | 16.2 (3.88)
  Total Change Score on RSES | 2.87 (3.42) | 0.20 (3.01)
Statistical Analysis 1: Comparison: Yoga Practice Group vs Attention Control Group; Statistical analysis examined Total Change Scores on RSES, using an independent samples t-test to evaluate null hypothesis that Total Change Score on RSES for each intervention group would be statistically comparable; Test type: Superiority or Other; p = 0.053, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected continuously over the 8 month period from recruitment to completion of all interventions (May 2010 through Jan 2011).
Groups:
- Yoga Practice Group: Participants in this group met for 90-minute sessions of hatha yoga practice twice a week for a total of 8 weeks. week for a total of 8 weeks.
- Attention Control Group: Participants in this group met for 90-minute education seminars on yoga history and philosophy twice a week for a total of 8 weeks.
Arm/Group | Yoga Practice Group | Attention Control Group
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/12
Other Adverse Events (participants affected / at risk) | 5/18 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yoga Practice Group (N=18) | Attention Control Group (N=12)
Musculoskeletal soreness or discomfort (Musculoskeletal and connective tissue disorders) | 5 (10) | 0 (0)

LIMITATIONS AND CAVEATS:
Small sample size; not possible to blind participants to intervention; sub-optimal adherence/completion rates, especially in attention control group; however, adherence/completion rates comparable to many exercise-based interventions for depression.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No